CLINICAL TRIAL: NCT01025687
Title: Effect of Television Viewing (TVV) & Puberty on Lunchtime Food Intake & Subjective Appetite in Girls
Brief Title: Television Viewing (TVV) & Puberty on Lunchtime Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: G. Harvey Anderson, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KidsStudy_21595
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Obesity Prevention
Keywords: girls; obesity; television viewing; puberty
MeSH Terms: conditions — Obesity | interventions — Water; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- glucose beverage (Experimental)
  Interventions: Dietary Supplement: water with glucose
- noncaloric beverage with TV (Experimental)
  Interventions: Behavioral: TV program showed while feeding
- glucose beverage with TV (Experimental)
  Interventions: Behavioral: TV program showed while feeding
- noncaloric beverage (Experimental)
  Interventions: Dietary Supplement: water with noncalorie sweetener

INTERVENTIONS:
Dietary Supplement: water with noncalorie sweetener
  Arms: noncaloric beverage
Dietary Supplement: water with glucose
  Arms: glucose beverage
Behavioral: TV program showed while feeding
  Arms: noncaloric beverage with TV
Behavioral: TV program showed while feeding
  Arms: glucose beverage with TV

SUMMARY:
The investigators hypothesize that television viewing will affect food intake in adolescent girls, and will depend on pubertal stage. Food intake will be measured at 30 min following a glucose(1 g of glucose/kg body weight) or sweetened noncaloric beverage with or without the presence of TV. Subjective appetite will be measured as well.

ELIGIBILITY:
Inclusion Criteria:

* healthy girls with no emotional, behavioral or learning problems

Exclusion Criteria:

* boys

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
food intake (kcal) | at 30 min after the treatment

SECONDARY OUTCOMES:
subjective appetite | 0-120 min

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, PhD., Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Patel BP, Bellissimo N, Thomas SG, Hamilton JK, Anderson GH. Television viewing at mealtime reduces caloric compensation in peripubertal, but not postpubertal, girls. Pediatr Res. 2011 Nov;70(5):513-7. doi: 10.1203/PDR.0b013e31822d783e. PMID 21772226